CLINICAL TRIAL: NCT03951506
Title: Effects a Multi-modal Exercise Program in Older Aduls With Knee Osteoarthritis
Brief Title: Multi-modal Exercise Program in Older Aduls With Knee Osteoarthritis
Acronym: MME-KOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-20
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-Multi-modal exercise program (Experimental): Each session (48) starts with 7 minutes of moderate warm-up exercises focusing on mobility and flexibility. Secondly, the strengthening exercises consist of knee extensions, knee flexions, hip abductions, ankle plantar flexions, and ankle dorsiflexions. Thirdly, a set of balance exercises including knee bends, backwards walking, walking and turning around, sideways walking, tandem stance, tandem walk,one-leg stand, heel walking, toe walking, toe to heel walking backwards, sit-to-stand, and stair walking. Finally, participants are instructed to walk at their usual pace for at least 10 minutes.
  Interventions: Other: Multi-modal exercise program
- Experimental-conventional treatment (Experimental): Each session (48) consist in isotonic exercises of low intensity and joint mobility of the lower extremities. These exercises are usually prescribed in medical consultations for the treatment of knee osteoarthritis.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Multi-modal exercise program — Each session (48) starts with 7 minutes of moderate warm-up exercises focusing on mobility and flexibility. Secondly, the strengthening exercises consist of knee extensions, knee flexions, hip abductions, ankle plantar flexions, and ankle dorsiflexions. Thirdly, a set of balance exercises including knee bends, backwards walking, walking and turning around, sideways walking, tandem stance, tandem walk,one-leg stand, heel walking, toe walking, toe to heel walking backwards, sit-to-stand, and stair walking. Finally, participants are instructed to walk at their usual pace for at least 10 minutes.
  Arms: Experimental-Multi-modal exercise program
Other: Conventional treatment — Each session (48) consist in isotonic exercises of low intensity and joint mobility of the lower extremities. These exercises are usually prescribed in medical consultations for the treatment of knee osteoarthritis.
  Arms: Experimental-conventional treatment

SUMMARY:
Aim: To evaluate the short-term effects of a multi-modal exercise program on physical performance variables in older adults with knee osteoarthritis.

DETAILED DESCRIPTION:
* Aim: To evaluate the short-term effects of 16 week multi-modal exercise program on physical performance variables in independent community-dwelling older adults with knee osteoarthritis.
* Design: randomized controlled trial.
* Setting: home-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Knee pain
* Score in Kellgren-Lawrence Scale ≥1

Exclusion Criteria:

* Unable to ambulate independently
* Mini-mental state examination score < 24
* Barthel Index score < 80
* Unstable cardiovascular disease
* Neurological disorder that could compromise exercising
* Upper or lower-extremity fracture in the past year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 16 weeks
  It is a self-questionnaire consisting of 24 items divided into 3 sub-scales: pain (5 items): when walking on level ground, using stairs, in bed, sitting or lying down, and standing. Rigidity (2 items) morning and during the rest of the day. Functional capacity (17 items): use of stairs, getting up from sitting, standing, stooping, walking, getting in / out of a car, going shopping, putting on / taking off socks and / or socks, getting out of bed, lying on the bed, entering / leaving the shower / tub, sitting and getting up from the toilet, performing heavy and light household chores.

SECONDARY OUTCOMES:
Numeric pain Rating Scale (NRS) | 16 weeks
  The NRS is a one-dimensional measure of pain intensity. The format is a line in which the participant selects a number between 0-10 that best reflects the intensity of the pain itself. A higher value corresponds to a greater intensity of pain.
Timed 10-Meter Walk Test (10-MWT) | 16 weeks
  It is a test for the evaluation of the usual and maximum gait speed along a distance of 10 meters corridor.
6-Minute Walk Test (6-MWT) | 16 weeks
  It is a test that evaluates the maximum distance a participant can walk during 6 minutes along a 30 meter long corridor.

CONTACTS AND LOCATIONS:
Overall Officials: JF Lisón, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided